CLINICAL TRIAL: NCT02304666
Title: Study of Inflammatory Markers (VNN1) in Crohn Disease and Ulcerative Colitis
Acronym: VANIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-33; 2014-A01237-40 (Other: Ansm)
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis)
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crohn disease's Patients (Experimental): Patients with Crohn disease or presenting an ulcerative colitis
  Interventions: Procedure: Colonoscopy for biopsies samples
- Control patient (Other): Patients with programmed colonoscopy screening for familial colon cancer history, polyps or for irritbale bowel syndrome
  Interventions: Procedure: Colonoscopy for biopsies samples

INTERVENTIONS:
Procedure: Colonoscopy for biopsies samples

SUMMARY:
Inflammatory Bowel diseases (IBD) include Crohn's disease and ulcerative colitis. IBD's precise origin is unknown until now. Today, the current hypothesis of the disease pathogenesis is that IBD result from a dysregulated mucosal immune response to the gut microbial flora in genetically susceptible hosts. The intestinal homeostasis depends on interactions between immune and epithelial cells. Epithelial cells are the first line of defense, are tightly connected to the underlying gut associated lymphoid tissue and their alteration results in loss of tissue homeostasis.

Vanin-1 (Vnn1 in mice, VNN1 in humans) is an epithelial pantheinase which regulates the cell response to stress.

This ectoenzyme hydrolyses the vitamin B5-derivative pantetheine to provide cysteamine to tissues and regenerate pantothenate. Previous studies have shown that Vnn1 KO mice were more resistant to experimental colitis and administration of cystamine (oxidized form of cysteamine) restored their susceptibility to colitis. Furthermore, analysis of VNN1 expression in IBD patients show that high VNN1 expression is associated with severe clinical features. Thus, analysis of VNN1 expression could represent a good prognostic marker.

In a recent published article, we characterized among a retrospective cohort of 500 IBD patients and controls new SNPs (single nucleotide polymorphisms) in the VNN1 promoter and showed their association with IBD incidence and high VNN1 expression. This suggested that the VNN1gene might be a new predisposition marker of IBD.

In mouse, Vnn1 expression is tightly regulated by activation of PPARa and PPARg transcription factors. Interestingly, one of the SNPs identified in patients participates to a PPARg binding site. Interestingly, drugs related to the family of 5-ASA which are commonly used in IBD, have PPARgamma agonist potential. Therefore, quantifying VNN1 levels in patients under 5-ASA therapy might help predicting response to therapy and select patients with the highest benefit for this therapy.

The purpose of this new project is to extend our initial analysis. The study will be prospective, monocentric and controlled. Its primary objective is to evaluate the level of VNN1 expression in the colonic mucosa between IBD patients and control subjects to confirm the correlation between high VNN1 expression and IBD. In relation with its prospective nature, we will also try to associate VNN1 expression level with specific endophenotypes (severity and/or localization of the lesions, quality of the response to therapy). Finally, we will screen patients for the previously identified SNPs to integrate this information in the interpretation of the results of expression analysis.

This study is planned on 2 years. Two groups of patients will be constituted: one group will include IBD patients followed in the " Service de Gastro-entérologie du Pr Grimaud à l'Hôpital Nord " and the other group will constitute the control cohort including persons who were proposed a screening colonoscopy for familial history of colon cancer or polyps, or for Irritable Bowel Syndrome.

The investigator will have to fill a questionnaire for each included patient, collecting information about age, sex, past medical history, taken medicine, digestive symptoms and colonoscopy indication.

IBD patients will have a first set of biopsies (n = 10) and blood samples collected under general anesthesia during a colonoscopy planned in their IBD usual follow-up; a second set of similar samples will be collected within the next 12 months if an endoscopic control is medically justified. The control subjects will have only one set of biopsy and blood samples collected under general anesthesia during their colonoscopy. In the particular case of IBD patients who require surgery, a small piece of the resection will be collected ex-vivo on both healthy and pathologic areas.

The blood sample will serve for quantification of the VNN1 seric pantheteinase activity and SNP's genetic study.

The colonic biopsies will be obtained in duplicates from 5 different ileocolonic areas, one for histopathological analysis and the other for transcriptional analysis by qRT-PCR.

The surgical samples will be used for transcriptional activity, tissue pantheteinase activity and constitution of TMA (Tissue MicroArrays) bank for immunohistochemistry.

Expected benefits are to validate a new IBD prognostic marker for disease severity or potentially for evaluation of the therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

Experimental group - Patients with Inflamatroy Bowel Disease

Control group:

-Patients that are planned to have a colonoscopy from familial history of colon cancer orpolyps or for irritable bowel syndroms

Both groups:

free informed consent signed

Exclusion Criteria:

* Patients with contradication for anesthesia
* Patient undergoind aspirin or anitinflamatory drugs within 72 hours of the colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Level of VNN1 expression | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France